CLINICAL TRIAL: NCT00737958
Title: The Effects of Diesel Exhaust Inhalation On Exercise Capacity In Patients With Stable Angina Pectoris
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Dr Jeremy Langrish, University of Edinburgh
Other Study IDs: BHF FS/07/048
Record Dates: First submitted 2008-08-19; First posted 2008-08-20 (Estimated); Last update posted 2010-03-31 (Estimated); Status verified 2008-07

CONDITIONS: Coronary Heart Disease; Angina Pectoris
Keywords: Angina pectoris; Air pollution; Diesel exhaust; Myocardial ischaemia; Exercise capacity
MeSH Terms: conditions — Coronary Disease; Angina Pectoris; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples Serum samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with documented stable coronary artery disease, symptoms of stable angina pectoris, and a positive standard BRUCE exercise stress test at 3 - 13 minutes.

SUMMARY:
The purpose of this study is to determine whether exposure to diesel exhaust (air pollution) has a functional impact on patients with stable angina pectoris.

DETAILED DESCRIPTION:
Air pollution is a major cause of cardiovascular morbidity and mortality. The mechanism and components of air pollution responsible for these cardiovascular effects are unknown but small combustion-derived particles are suspected to be the major cause. Using a unique exposure system in Umeå Sweden, we have demonstrated that healthy volunteers who inhale dilute diesel exhaust develop an impairment of two important, highly relevant and complementary aspects of vascular function: the regulation of vascular tone and endogenous fibrinolysis. We have recently extended these findings and have shown that brief exposure to dilute diesel exhaust promotes myocardial ischemia and inhibits endogenous fibrinolytic capacity in patients with stable asymptomatic coronary heart disease. We now wish to extend these findings to patients with chronic stable angina pectoris. In particular, we wish to determine the functional impact of diesel exhaust inhalation as well as describe the time course and minimum exposure that can induce these detrimental effects.

ELIGIBILITY:
Inclusion Criteria:

* Documented coronary heart disease
* Symptoms of stable angina pectoris

Exclusion Criteria:

* History of arrhythmia
* Severe 3 vessel coronary artery disease or left main stem stenosis that has not been revascularised
* Resting conduction abnormality
* Digoxin therapy
* Uncontrolled hypertension
* Renal or hepatic failure
* Patients with unstable disease (ACS or unstable symptoms within 3 months)
* Asthma
* Intercurrent illness

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be recruited from the cardiology outpatient clinics
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2008-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Myocardial ischaemia - measured as time to 1mm ST segment depression on the ECG during standard BRUCE exercise stress testing. | Immediately after exposure

SECONDARY OUTCOMES:
Total ischaemic burden - assessed using 24 hour Holter ambulatory ECG monitoring | 24hrs after exposure
Total exercise capacity - assessed by maximal work done during exercise stress test | Immediately after exposure
Biochemical evidence of myocardial ischaemia - plasma highly sensitive troponins, ischaemically modified albumin, fatty acid binding protein | Before, after and at 24 hours after exposure

CONTACTS AND LOCATIONS:
Overall Officials: David E Newby, MD FRCP, Study Director — University of Edinburgh
Locations (1):
- University of Edinburgh, Edinburgh, Midlothian, United Kingdom

REFERENCES:
- [Background] Mills NL, Tornqvist H, Gonzalez MC, Vink E, Robinson SD, Soderberg S, Boon NA, Donaldson K, Sandstrom T, Blomberg A, Newby DE. Ischemic and thrombotic effects of dilute diesel-exhaust inhalation in men with coronary heart disease. N Engl J Med. 2007 Sep 13;357(11):1075-82. doi: 10.1056/NEJMoa066314. PMID 17855668
- [Background] Tornqvist H, Mills NL, Gonzalez M, Miller MR, Robinson SD, Megson IL, Macnee W, Donaldson K, Soderberg S, Newby DE, Sandstrom T, Blomberg A. Persistent endothelial dysfunction in humans after diesel exhaust inhalation. Am J Respir Crit Care Med. 2007 Aug 15;176(4):395-400. doi: 10.1164/rccm.200606-872OC. Epub 2007 Apr 19. PMID 17446340
- [Background] Mills NL, Tornqvist H, Robinson SD, Gonzalez M, Darnley K, MacNee W, Boon NA, Donaldson K, Blomberg A, Sandstrom T, Newby DE. Diesel exhaust inhalation causes vascular dysfunction and impaired endogenous fibrinolysis. Circulation. 2005 Dec 20;112(25):3930-6. doi: 10.1161/CIRCULATIONAHA.105.588962. PMID 16365212
- [Background] Lanki T, Hoek G, Timonen KL, Peters A, Tiittanen P, Vanninen E, Pekkanen J. Hourly variation in fine particle exposure is associated with transiently increased risk of ST segment depression. Occup Environ Med. 2008 Nov;65(11):782-6. doi: 10.1136/oem.2007.037531. Epub 2008 Jun 4. PMID 18524840
- [Background] Pekkanen J, Peters A, Hoek G, Tiittanen P, Brunekreef B, de Hartog J, Heinrich J, Ibald-Mulli A, Kreyling WG, Lanki T, Timonen KL, Vanninen E. Particulate air pollution and risk of ST-segment depression during repeated submaximal exercise tests among subjects with coronary heart disease: the Exposure and Risk Assessment for Fine and Ultrafine Particles in Ambient Air (ULTRA) study. Circulation. 2002 Aug 20;106(8):933-8. doi: 10.1161/01.cir.0000027561.41736.3c. PMID 12186796